CLINICAL TRIAL: NCT05124613
Title: The Impact of Covid-19 on Patients Waiting for Elective Knee Surgery: An Investigation Into Patient Perceptions of Knee Function and Pain
Brief Title: The Impact of Covid-19 on Patients Waiting for Knee Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Leela Biant, Professor, University of Manchester
Other Study IDs: NHS001829
Record Dates: First submitted 2021-03-06; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee; Osteochondral Defect; Cartilage Injury; Cartilage Damage; Knee Injuries; Knee Injuries and Disorders
Keywords: COVID-19; Knee Surgery; Knee Pain; Knee Function; Coping Mechanisms
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries; Disease; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients waitlisted for Knee Surgery: Adults identified by a consultant orthopaedic surgeon at the study site as being on a waiting list for surgery on their knee and as experiencing a delay to their knee surgery as a result of the COVID-19 pandemic will be eligible to participate in this survey. The survey will include one validated questionnaire and a series of bespoke questions.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Information collected and stored in Survey:
  * Type of knee surgery the patient is waitlisted for
  * Demographics: age, sex, recent weight gain
  * Validated and bespoke questions:
    1. EQ-5D survey (a validated questionnaire on health)
    2. Bespoke questions on knee pain today
    3. Bespoke questions on knee function today
    4. Bespoke questions on change in knee pain since being waitlisted for surgery
    5. Bespoke questions on change in knee function since being waitlisted for surgery
    6. Bespoke questions on coping mechanisms patients use to manage symptoms
    7. Bespoke questions on what support they would find beneficial whilst they wait for their surgery
    8. Three bespoke questions about COVID-19 (Have they ever tested positive/Has the pandemic changed their mind about wanting surgery/Has the perception of their knee pain and function changed since the first lockdown was introduced?)

SUMMARY:
The Covid-19 pandemic has led to the postponement and cancellation of elective orthopaedic surgeries worldwide. These delays to elective procedures combined with ongoing demand have led to increasingly longer waiting list times.

This cross-sectional pilot study aims to investigate the change in patients' perceptions of knee pain and function since being waitlisted for surgery. A bespoke survey will be administered to eligible patients over the phone from Trafford General Hospital, Manchester. The survey will also investigate the coping mechanisms and the preventative measures patients are taking to manage symptoms during the pandemic, and question what kinds of communication and support patient would like to be offered whilst waiting for treatment.

This study will improve clinicians' and researchers' understanding of how patients are coping with symptoms during this pandemic, and provide information on how to better support patients who are waiting for knee surgery. This information could be used to enhance orthopaedic care during, and in the aftermath, of this pandemic. The information gathered in this study may also be used to inform a larger multi-centre study.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified by a consultant orthopaedic surgeon as being on a waiting list for surgery on their knee.
* Patients identified by a consultant orthopaedic surgeon who are experiencing a delay to their knee surgery as a result of the COVID-19 pandemic.
* Patients over 18 years old.

Exclusion Criteria:

* Patients who are no longer waiting for their surgery (e.g. surgery performed elsewhere or patient has changed their mind about undergoing surgery).
* Patients who are on a waiting list for any surgery other than surgery of the knee.
* Patients who are on a waiting list for surgery at a hospital which is not a part of Manchester University NHS Foundation Trust.
* Patients who cannot read and speak English.
* Patients who cannot complete the survey over the phone.
* Patients who cannot give informed consent due to cognitive impairment (e.g. dementia or similar cognitive condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults awaiting surgery on the knee who have experienced delays to their procedure due to the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in perceived knee pain | Up to 2 years
  The survey will ask patients to compare the level of pain they have in their knee now to the level of pain they had in their knee when they were put on the waiting list for knee surgery
Change in perceived knee function | Up to 2 years
  The survey will ask patients to compare the level of function they have in their knee now to the level of function they had in their knee when they were put on the waiting list for knee surgery

SECONDARY OUTCOMES:
Change in symptom management | Up to 2 years
  The survey will ask patients to describe how they are managing their symptoms during the COVID-19 pandemic and describe whether this has changed since the pandemic started.
Support | Up to 1 year
  The survey will ask patients to describe what kinds of support they would like to receive whilst they wait for their delayed surgery to take place (current).

CONTACTS AND LOCATIONS:
Locations (1):
- Trafford General Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers.